CLINICAL TRIAL: NCT03386084
Title: Efficacy of Motor Control Treatment Combined With Resistive Capacitive Diathermy in Acute Low Back Pain
Brief Title: Efficacy of Motor Control and Diathermy Treatment in Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, MIGUEL ANGEL CAÑADAS GARCIA, Physiotherapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM/HU/2017/19
Record Dates: First submitted 2017-11-29; First posted 2017-12-29 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Low Back Pain
Keywords: capacitive resistive diathermy; motor control
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct application of microwave diathermy and motor control (Experimental)
  Interventions: Device: microwave diathermy
- application of microwave diathermy without therapeutic effects (Placebo Comparator)
  Interventions: Device: microwave diathermy

INTERVENTIONS:
Device: microwave diathermy — Application of microwave diathermy with Monopolar CapacitiveResistive Radiofrequency Therapy (INDIBA)

SUMMARY:
Lumbar pain is considered one of the most frequent health problems faced by human populations on a global scale.

This study will be carried out to evaluate the efficiency of motor control treatments combined with diathermy in patients diagnosed with acute lower back pain, focusing upon the potential for accelerated patient recuperation if both treatments are applied simultaneously and jointly.

ELIGIBILITY:
Inclusion Criteria:

* Acute low back pain (no more of 4 weeks)
* Spanish speaker
* Between 18-65 years

Exclusion Criteria:

* Patients in whom diathermy is a contraindicated therapy
* Pacemaker
* Pregnant
* Not intact skin
* Thrombophlebitis
* Hypotension
* Anticoagulated patient or with local surgical intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Pain | 4 weeks
  An unpleasant sensation induced by noxious stimuli which are detected by nerve endings of nociceptive neurons.
  The measurement tool that will be used is Visual Analog Scale. This scale is a unidimensional measure of pain intensity. It has a continuous scale comprised of a horizontal line with an interval of 10 points, where 1 is the minimum intensity of pain the patient can endure and 10 is the maximum intensity of pain the patient can endure.

SECONDARY OUTCOMES:
Disability | 4 weeks
  Determination of the degree of a physical patient´s handicap. The measurement tool that will be used is Roland Morris Disability Questionnaire. This questionnaire is used to establish physical disability degree of people with non specific acute low back pain. It has 24 questions the patient should point out to determinate his/her limitation for make normal activities.
Satisfaction | 4 weeks
  To evaluate the assessment of the satisfaction regarding the attention and quality of the services received and the degree of compliance with the patient's expectations about the treatment.
  The measurement tool that will be used is Client Satisfaction Questionnaire. This questionnaire is used to evaluate patient's satisfaction with the care and quality of the health services received. It has 8 items from 1 to 4 points (where 1 is the minimum satisfaction and 4 is the maximum satisfaction) to assess the satisfaction degree.

CONTACTS AND LOCATIONS:
Locations (1):
- FisioWork, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided